CLINICAL TRIAL: NCT00002749
Title: PHASE II STUDY OF CARBOPLATIN (CBDCA) IN THE TREATMENT OF CHILDREN AND ADULTS WITH PROGRESSIVE LOW GRADE GLIOMAS
Brief Title: Carboplatin in Patients With Progressive Gliomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Henry Friedman, MD, Duke UMC
Purpose: Treatment
Other Study IDs: CDR0000064682; DUMC-0157-00-1R7; DUMC-0137-99-1R6; DUMC-081-96-1R3; DUMC-115-97-1R4; DUMC-118-98-1R5; NCI-V96-0868
Record Dates: First submitted 1999-11-01; First posted 2004-08-11 (Estimated); Last update posted 2009-10-14 (Estimated); Status verified 2009-10

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: childhood low-grade cerebral astrocytoma; recurrent adult brain tumor; adult brain stem glioma; childhood oligodendroglioma; untreated childhood brain stem glioma; recurrent childhood brain stem glioma; untreated childhood visual pathway glioma; recurrent childhood visual pathway glioma; untreated childhood cerebellar astrocytoma; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; adult anaplastic astrocytoma; adult oligodendroglioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Oligodendroglioma; Optic Nerve Glioma; Astrocytoma | interventions — Carboplatin

INTERVENTIONS:
Drug: carboplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of carboplatin in patients with progressive glioma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the response to carboplatin (CBDCA) in patients with progressive low-grade gliomas. II. Assess the activity of CBDCA in stabilizing the growth of these tumors.

OUTLINE: Single-Agent Chemotherapy. Carboplatin, CBDCA, NSC-241240.

PROJECTED ACCRUAL: A total of 25 evaluable patients will be entered if there is at least 1 response in the first 9 patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed primary intracranial low-grade glioma (i.e., astrocytoma or oligodendroglioma) No more than 2 years since tissue diagnosis Biopsy not required for intrinsic chiasmatic mass or tumor infiltration along the posterior optic tracts Evidence of progressive disease by at least one of the following: Papilledema or other clinical sign of increased intracranial pressure Documented change in neuroimaging studies, e.g.: Hydrocephalus 25% increase in product of maximum perpendicular diameters of tumor The following are required in patients with optic pathway gliomas: Progressive loss of vision documented by an ophthalmologist, i.e.: Doubling of octaves (e.g., 20/20 to 20/40 or 20/40 to 20/80) on 2 successive visits Loss of visual acuity not explainable by other causes, e.g., media abnormalities or amblyopia Greater than 3 mm increase in proptosis At least 2 mm increase in diameter of optic nerve on neuroimaging Increase in distribution of tumor involving the optic tracts or optic radiations demonstrated by CT or MRI using T1 (with or without contrast) or T2 imaging

PATIENT CHARACTERISTICS: Age: Any age Performance status: Karnofsky 70%-100% Life expectancy: At least 12 weeks Hematopoietic: ANC at least 1,500 Platelets at least 100,000 Hemoglobin at least 8.0 g/dL Hepatic: Bilirubin less than 1.5 times normal ALT less than 1.5 times normal Renal: Creatinine less than 1.5 mg/dL Other: Negative pregnancy test required of fertile women Effective contraception required of fertile patients

PRIOR CONCURRENT THERAPY: At least 12 weeks since radiotherapy (4 weeks since other therapy) and recovered Prior chemotherapy allowed with subsequent disease progression

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 1993-02; Study Completion 2000-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry S. Friedman, MD, Study Chair — Duke University
Locations (2):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States
- Hopital Sainte Justine, Montreal, Quebec, Canada